CLINICAL TRIAL: NCT01712581
Title: Determination of Myocardial Relaxation Times Values in Healthy Volunters
Brief Title: Heart Map Study -Determination of Myocardial Relaxation Times Values in Healthy Volunters
Acronym: HeartMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/071/HP
Record Dates: First submitted 2012-10-17; First posted 2012-10-23 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Normal Myocardial T1, T2 and T2* Values
Keywords: normal myocardial T1, T2 and T2* values
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy volunters (Experimental): 175 Healthy volunters in the cohorte divided in 7 groups of age: 18-19 years old (ratio M/F: 1/1) 20-24 years old (ratio M/F: 1/1) 25-29 years old (ratio M/F: 1/1) 30-39 years old (ratio M/F: 1/1) 40-49 years old (ratio M/F: 1/1) 50-59 years old (ratio M/F: 1/1) 60-69 years old (ratio M/F: 1/1)
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging

SUMMARY:
T1, T2 and T2* relaxation times, as determined with cardiac MRI, are markers of myocardial tissue content (water, fibrosis, iron).

The aim of study is to determine the normal values of T1, T2 and T2* relaxation times in healthy volunters aged 18-69 years using 1.5T clinical MRI.

DETAILED DESCRIPTION:
Cardiac MRI is more and more used in patients with ischaemic and non-ischaemic heart diseases. One major strength of MRI is its great potential for tissue characterization.

For early detection and follow-up of patients with hemosiderosis, who are at high risk of myocardial iron overload, cardiac MRI seems to be the most reliable, more reproducible and less invasive method. In addition MRI does not require injection of contrast media. It is commonly accepted that myocardial T2 * value of less than 20 ms corresponds to iron overload in the myocardium. However, this value is based on a small sample study and nomogram based on age were not published. The determination of normal values in a population of healthy controls according to age appears to be a prerequisite for reliable interpretation of imaging data.

Moreover, myocardial edema and fibrosis are more and more evaluated with cardiac MRI using T1 and T2 myocardial relaxation times. As for T2* values, normogram of T1 and T2 values based on age were not published.

The increasing use of T1, T2 and T2* mapping sequences in clinical practice for tissue characterization of the myocardium justify the implementation of a study in healthy volunteers to determine normograms based on age.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers over the age of 18 and less than 70
* Volunteers able to understand and sign the consent and to give written informed consent
* Female contraceptives if of childbearing age
* Registered or entitled to social security system
* Volunteers able to maintain supine for 20 minutes

Exclusion Criteria:

* Major protected/under guardianship
* Volunteers unable to maintain the supine position for 20 minutes
* Claustrophobia
* Volunteers with history of PRBC transfusion
* Volunteers with history of hematologic disease or a disruption of iron status
* Volunteers with history of cardiac disease including arrhythmias
* Hypertension
* Diabetes
* Contra-indication for MRI: metal fragments in the eyes; implantable cardiac, neurological or ENT device; osteosynhesis material not compatible with MRI
* Women who are pregnant or likely to be

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The main objective is to determine normal T2 * values of the myocardium in a large adult population of healthy volunteers, using 1.5T cardiac MRI. | 24h

SECONDARY OUTCOMES:
The secondary objectives are to determine normal T1 and T2 values of the myocardium in a large adult population of healthy volunteers, using 1.5T cardiac MRI. | 24h

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France